CLINICAL TRIAL: NCT04170972
Title: The Role of TBC1D4 in Exercise- and Insulin-induced Glucose Metabolism in Human Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Professor Jorgen FP Wojtaszewski, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KVUG 2016-12; H-18007316 (Other: The Danish National Committee on Health Research Ethics); 13057 (Other Grant/Funding Number: Novo Nordisk Foundation); 5053-00095B (Other Grant/Funding Number: Danish Council for Independent Research); 28136 (Other Grant/Funding Number: Steno Collaborative Grant)
Record Dates: First submitted 2019-04-23; First posted 2019-11-20 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-04

CONDITIONS: Exercise; Insulin Sensitivity; Skeletal Muscle
MeSH Terms: conditions — Motor Activity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A case-control study with two groups of participants with different genetic background on the TBC1D4 gene:
  1. Homozygote carriers of a p.Arg684T TBC1D4 gene-variant
  2. None carriers (matched controls) of the p.Arg684T TBC1D4 gene-variant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and vivo insulin stimulation in TBC1D4 gene-variants (Experimental): Acute exercise and in vivo insulin stimulation in homozygote carriers of a p.ARg684T TBC1D4 gene-variant.
  Interventions: Other: Acute exercise
- Exercise and vivo insulin stimulation in matched controls (Experimental): Acute exercise and in vivo stimulation in none carriers (matched controls) of the p.Arg684T TBC1D4 gene-variant.
  Interventions: Other: Acute exercise

INTERVENTIONS:
Other: Acute exercise — One hour of acute one-legged knee-extensor exercise followed by 3 hours recovery and 2 hours insulin (1.5 mU/min/kg) stimulation.
  Other Names: Insulin stimulation

SUMMARY:
Recently a common Greenlandic nonsense p.Arg684erTer variant (in which arginine is replaced by a termination codon) in the gene TBC1D4 was discovered. The variant has an allele frequency of 17%. Homozygous carriers of this TBC1D4 variant have impaired glucose tolerance and a 10-fold enhanced risk of developing type 2 diabetes (T2D). The investigators propose to carry out comprehensive metabolic phenotyping of adult Inuits carrying zero or two alleles of the TBC1D4 variant. The investigators hypothesise that regulation of TBC1D4 in skeletal muscle is pivotal in regulating glucose uptake during exercise, during physiological insulin stimulation, and for the ability of an acute bout of exercise to improve insulin sensitivity to regulate glucose metabolism in humans.

The overall aims in the present project are to:

1. Determine whether the TBC1D4 p.Arg684Ter variant affects the regulation of glucose uptake in skeletal muscle during exercise and during physiological insulin stimulation.
2. Determine the effect of the TBC1D4 p.Arg684Ter variant for the ability of acute exercise to insulin sensitize skeletal muscle to regulate glucose metabolism.
3. Define the metabolic pathways affected by the p.Arg684Ter variant in order to identify causal factors responsible for the diabetic phenotype of Inuit carriers.

The knowledge generated will contribute to additional explanatory clues to the increased frequency of T2D in the carriers.

DETAILED DESCRIPTION:
Recently a common Greenlandic nonsense p.Arg684erTer variant (in which arginine is replaced by a termination codon) in the gene TBC1D4 was discovered. The variant has an allele frequency of 17%. Homozygous carriers of this TBC1D4 variant have impaired glucose tolerance and a 10-fold enhanced risk of T2D. The investigators propose to carry out comprehensive metabolic phenotyping of adult Inuits carrying zero or two alleles of the TBC1D4 variant. The investigators hypothesise that regulation of TBC1D4 in skeletal muscle is pivotal in regulating glucose uptake during exercise, during physiological insulin stimulation, and for the ability of an acute bout of exercise to improve insulin sensitivity to regulate glucose metabolism in humans.

Our overall aims in the present project are to:

1. Determine whether the TBC1D4 p.Arg684Ter variant affects the regulation of glucose uptake in skeletal muscle during exercise and during physiological insulin stimulation.
2. Determine the effect of the TBC1D4 p.Arg684Ter variant for the ability of acute exercise to insulin sensitize skeletal muscle to regulate glucose metabolism.
3. Define the metabolic pathways affected by the p.Arg684Ter variant in order to identify causal factors responsible for the diabetic phenotype of Inuit carriers.

The knowledge generated will contribute to additional explanatory clues to the increased frequency of T2D in the carriers.

Study population:

The Inuit Health in Transition (IHIT) study is a study of adults in West and East Greenland. The participants were selected through a stratified random sample and data were collected in 1999-2010 using clinical procedures, sampling of biological material, and questionnaires. To accomplish the goal, the investigators will carry out comprehensive metabolic phenotyping of Inuits carrying zero (n=10) or two (n=10) alleles of the TBC1D4 p.Arg684Ter variant recruited from this cohort. Based on an effect of 1.2 SD as found for plasma glucose levels during an Oral Glucose Tolerance Test (OGTT) in the previous study (6) between homozygous carriers and non-carriers of the TBCD14 variant, the investigators achieve 89% power at p=0.05 when recruiting 10 homozygous carriers and 10 non-carriers.

Methods:

Genotyping of the IHIT cohort has already been performed. Thus, the investigators can re-call study participants for the present study based on their known genotype. The investigators intend to perform highly invasive physiological studies of subjects harboring the TBC1D4 point mutation and in control subjects matched by age, gender and BMI. The participants will be nondiabetic (25-50 yrs) males recruited through the IHIT cohort register (n=4,200). The recruitment, screening and initial clinical investigations (oral glucose tolerance test and physical exercise tests, including customization to a one-legged cycling ergometer) will take place in Greenland. The most invasive part of the study, described below, will take place in Copenhagen, Denmark.

During the stay in Copenhagen participants will receive an energy-matched, standardized diet to be consumed 3 days prior to the intervention study. On the study day the participants will arrive in the laboratory after an overnight fast. Catheters will be placed in both femoral veins (V) and in one femoral artery (A). A muscle biopsy will be obtained from vastus lateralis of one leg (resting leg). The participants will then perform one legged knee extensor exercise for one hour leaving the other leg as a rested control leg. Immediately after exercise a biopsy will be obtained from the exercising leg and the participants will rest in the fasted state for 3 hours before a third set of muscle biopsies (from both legs) and one abdominal subcutaneous fat biopsy are taken. Subsequently, insulin sensitivity will be evaluated during a 2-hour physiological hyperinsulinemic euglycemic clamp. By the end of the clamp a final set of biopsies (both legs) and one abdominal subcutaneous fat biopsy will be obtained. Throughout the study day sampling of artery and venous blood/plasma samples allow estimation of substrate extraction by the two legs. Further, measures of artery blood flow by Ultrasound Doppler technique will allow a final calculation of substrate uptake/release across the two legs before exercise, during exercise and in recovery from exercise. Importantly, the ability for insulin to stimulate theses process can be evaluated in both a rested and in the prior exercised leg.

The investigators plan to carry out deep transcript profiling of muscle tissue samples and define correlations between age, sex, BMI, genetic variants, and the transcriptional profiles in order to understand the impact on gene regulation of identified metabolic genetic variants. In order to define key biochemical pathways affected by the mutated TBC1D4, the investigators will perform metabolomic analyses of the muscle biopsy samples. In order to identify putative targeted pathways affected by the mutation, the investigators will perform mass spectrometry-based interactome as well as proteomic / phosphoproteomic analyses. Based on these data and data obtained from the metabolic analyses, the investigators will be better able to identify the affected metabolic processes involved in the progression towards the diabetic phenotype of the Inuit carriers. Such pathways will in subsequent analyses be studied biochemically in more detail including additional (to phosphorylation) post translational modifications (e.g. glycosylation) as well as expression/activities of key enzymes in glucose and fat metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Homozygote carriers of a pArg684T gene-variant (cases) and matched non carriers (controls)
* BMI between 20-35 kg/m2

Exclusion Criteria:

* Medical treated type 2 diabetes patients

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in leg glucose uptake | Measured 14 times during the experimental day (dispersed over 6 hours)
  Leg glucose uptake is calculated by the arterial-venous difference i blood glucose concentration multiplied with leg blood flow. Sampling of artery and venous blood samples for blood glucose measurements. Measures of artery blood flow by Ultrasound Doppler technique allows a final calculation of glucose uptake across the legs before exercise, during exercise, in recovery from exercise and with insulin stimulation.
Changes in whole body insulin sensitivity sensitivity. | 6 times (each 20 minutes) during 2 hours insulin stimulation.
  Insulin stimulated glucose uptake at whole body level (glucose infusion rate)
Metabolome. | At 4 times points: Before exercise, immediately after exercise, 3 hours after exercise and after 2 hours of insulin stimulation.
  Metabolomic analyses to map changes in biochemical pathways in skeletal muscle.
Transcriptome. | At 4 times points: Before exercise, immediately after exercise, 3 hours after exercise and after 2 hours of insulin stimulation.
  Transcriptome sequencing in skeletal muscle.
Changes in the TBC1D4 interactome. | At 4 times points: Before exercise, immediately after exercise, 3 hours after exercise and after 2 hours of insulin stimulation.
  TBC1D4 interactome analyses, to identify TBC1D4 signaling partners
Proteome and phosphoproteome. | At 4 times points: Before exercise, immediately after exercise, 3 hours after exercise and after 2 hours of insulin stimulation.
  Proteomics and targeted phosphoproteomic to identify changes in skeletal muscle.
Changes in phosphorylation and glycosylation signatures of TBC1D4 | At 4 times points: Before exercise, immediately after exercise, 3 hours after exercise and after 2 hours of insulin stimulation.
  Phosphorylation and glycosylation signatures of the TBC1D4 protein by western blotting to describe regulation of TBC1D4.
Changes of canonical intermediates in insulin- and exercise-induced signaling | At 4 times points: Before exercise, immediately after exercise, 3 hours after exercise and after 2 hours of insulin stimulation.
  Expression and/or activity of canonical intermediates in insulin- and exercise-induced signaling and metabolic pathways.
Changes in leg substrate utilization | At 4 times points: Before exercise, immediately after exercise, 3 hours after exercise and after 2 hours of insulin stimulation.
  Throughout the study day sampling of artery and venous blood/plasma samples allow estimation of substrate utilization based on the respiratory quotient (RQ).

SECONDARY OUTCOMES:
Substrate metabolism in primary myotubes from TBC1D4 p.Arg684 variant carriers and controls | At two conditions: With and without insulin.
  Mechanistic in vitro studies of the TBC1D4 p.Arg684 variant on glucose and fat metabolism.
Activities of key enzymes in glucose and fat metabolism | at 2 time points: Before and after 2 hours of insulin stimulation.
  Expression/activities of key enzymes in glucose and fat metabolism in adipose tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Exercise, Nutrition and Sports, Faculty of Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moltke I, Grarup N, Jorgensen ME, Bjerregaard P, Treebak JT, Fumagalli M, Korneliussen TS, Andersen MA, Nielsen TS, Krarup NT, Gjesing AP, Zierath JR, Linneberg A, Wu X, Sun G, Jin X, Al-Aama J, Wang J, Borch-Johnsen K, Pedersen O, Nielsen R, Albrechtsen A, Hansen T. A common Greenlandic TBC1D4 variant confers muscle insulin resistance and type 2 diabetes. Nature. 2014 Aug 14;512(7513):190-3. doi: 10.1038/nature13425. Epub 2014 Jun 18. PMID 25043022